CLINICAL TRIAL: NCT07253870
Title: Comparative Effects of Transcutaneous Auricular and Cervical Vagus Nerve Stimulation on Upper Limb Function, Cognition and Quality of Life in Subacute Stroke Patients
Brief Title: Comperative Effects of Transcutaneous Auricular and Cervical Vagus Nerve Stimulation in Subacute Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/O32 Wafa
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Stroke, Acute
Keywords: Task Specific Training; Upper Limb Function; Cognition
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Interventional study model for this study is a parallel-group randomized clinical trial (RCT). This model involves two distinct groups:
  Treatment Group A Participants will receive transcutaneous vagus nerve stimulation through auricular branch along with task specific exercises Treatment Group B Participants will receive transcutaneous vagus nerve stimulation through cevical branch along with task specific exercises Each participant is assigned randomly to one of these groups, ensuring that comparisons between the groups is unbiased. This parallel structure means each group undergoes its specific intervention throughout the study period without crossover to the other group's intervention. This approach helps assess the suitable tVNS approach for improving functional independence and quality of life for stroke survivors
Who Masked: Participant, Outcomes Assessor
Masking Description: outcome assessor will be blind about participants allocation. this will ensure that their evaluations are objective and not influenced by knowledge of which treatment group participants belong to. Participants in both groups will be masked to the treatment of the other group by scheduling their sessions at different times.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous vagus nerve stimulation through auricular branch along with task specific exercises (Experimental): Group A will receive application of TENS to stimulate the vagus nerve at the ear level, apply the clip electrodes at the targus/cymba concha and the other electrode anywhere in the skin over neck along with task specific exercises
  Interventions: Other: Transcutaneous vagus nerve stimulation through auricular branch along with task specific exercises
- Transcutaneous vagus nerve stimulation through cervical branch along with task specific exercises (Active Comparator): Group B will receive application of TENS to stimulate the vagus nerve at the neck level, apply the pad electrodes at the anterior mid to neck and the other electrode over back of neck along task specific exercises
  Interventions: Other: Transcutaneous vagus nerve stimulation through cervical branch along with task specific exercises

INTERVENTIONS:
Other: Transcutaneous vagus nerve stimulation through auricular branch along with task specific exercises — Group A will receive application of TENS to stimulate the vagus nerve at the ear level, apply the clip electrodes at the targus/cymba concha and the other electrode anywhere in the skin over neck Mode on TENS will be normal, with the width pulse of 250µs. FITT will be as follow Frequency of 25 Hz, Intensity 1mA, Time 30 minutes and the treatment will be of 5 days a week for 8 consecutive weeks
  * For grip and release: Use a soft ball, putty, or other textured objects. The patient squeezes the object to strengthen their grip and then releases it.
  * Reaching task: Place objects at varying distances in front of the patient. Encourage them to reach out with the affected arm to grasp the items and then bring them back.
  * Bilateral arm movement: Encourage simultaneous reaching or moving with both arms (e.g., pushing against a wall or lifting a lightweight object) to promote symmetry and coordination. Improve coordination and function of both arms.
  * Tabletop activities: Engaging in activities lik
  Arms: Transcutaneous vagus nerve stimulation through auricular branch along with task specific exercises
Other: Transcutaneous vagus nerve stimulation through cervical branch along with task specific exercises — Group B will receive application of TENS to stimulate the vagus nerve at the neck level, apply the pad electrodes at the anterior mid to neck and the other electrode over back of neck Mode on TENS will be normal, with the width pulse of 250µs. FITT will be as follow Frequency of 25 Hz, Intensity 1mA, Time 30 minutes and the treatment will be of 5 days a week for 8 consecutive weeks
  * For grip and release: Use a soft ball, putty, or other textured objects. The patient squeezes the object to strengthen their grip and then releases it.
  * Reaching task: Place objects at varying distances in front of the patient. Encourage them to reach out with the affected arm to grasp the items and then bring them back.
  * Bilateral arm movement: Encourage simultaneous reaching or moving with both arms (e.g., pushing against a wall or lifting a lightweight object) to promote symmetry and coordination. Improve coordination and function of both arms.
  * Tabletop activities: Engaging in activities like sortin
  Arms: Transcutaneous vagus nerve stimulation through cervical branch along with task specific exercises

SUMMARY:
This study aims to determine whether transcutaneous vagus nerve stimulation (tVNS) via auricular or cervical branches enhances recovery when combined with task-specific training in subacute stroke patients. We anticipate finding that both stimulation methods may improve upper limb motor function compared to conventional therapy. The research is expected to reveal specific cognitive domains (attention, memory, executive function) that benefit most from each stimulation approach, while also demonstrating meaningful improvements in patients' quality of life measures. These findings may make a significant practical contribution by providing clinicians with evidence-based guidance on suitable tVNS approach for improving functional independence and quality of life for stroke survivors.

DETAILED DESCRIPTION:
Stroke is characterized as a neurological deficit resulting from a sudden focal injury to central nervous system due to vascular issue by blockage and rupture of artery that leads to hypoxic injury and ultimately cell death. Stroke is primarily categories into two types: ischemic stroke that accounts for 85 % of cases and haemorrhagic stroke which make up 15%. Stroke leads to physical, cognitive, speech, perceptual and psychological Impairments. Post stroke impairments of the upper limb and lower limb leads to activity limitations in self-care and mobility and restricted participation in caring family and employment.

Multidisciplinary approach is used in stroke rehabilitation to create a rehabilitation program that aim to improve the function and improve the quality of life. Physical medicine and rehabilitation is focused on promoting recovery, improving or restoring functional abilities, anticipating potential long-term complications, and enhancing the quality of life for individuals with physical impairments or disabilities. Now a days there are many contemporary approaches used in rehabilitation like non-invasive brain simulation, robotics, gamification, virtual reality, CIMT, mirror therapy and many others, aimed to enhance the recovery after stroke.

Transcutaneous vagus nerve stimulation tVNS was developed two decades ago as a non-invasive, cost effective and easily applicable treatment option as compared to invasive vagus nerve stimulation for the treatment of epilepsy, cognitive impairments and stroke rehabilitation. Cutaneous innervation of vagus nerve is by two branches, one through auricular branch at external acoustic meatus, inner tragus, and the periauricular skin surrounding the cymba conchae and the other through cervical branch at anterior to sternocleidomastoid at the mid of neck. Several devices are used for stimulating the vagus nerve transcutaneously, as NEMOS that stimulates at the concha of outer ear, CE (European Conformity) and a hand held device Gammacore. On the other hand TENS-200 or Digitimer DS7A often require custom-made electrodes, also used in stimulation. In 2018 a systematic review was conducted on the safety of tVNS that results in transcutaneous vagus nerve stimulation (tVNS) is generally well tolerated in humans at the tested doses and is considered safe.

In parasympathetic nervous system vagus nerve is a major component that emerges from the medullae oblongata, passes through the jugular foramen to leave the cranial activity and travel downward between the neurovascular bundle situated between internal jugular vein and common carotid artery. It extends to thoracic and abdominal cavities and supply multiple organs and regulate autonomic nervous system. VNS play its role by stimulating the afferent and efferent fibers of the VN that primarily comprises the unmyelinated sensory afferent fibers, accounting for 80-90% of the nerve fiber, with the remaining 10-20% being myelinated efferent fibers. These fibers project upward to the brainstem nucleus and relay circuit, influencing the nucleus tractus solitarius (NTS) and locus coeruleus (LC). NTS projects different brain areas as amygdala, hippocampus, locus coeruleus and prefrontal cortex. The effects of direct VNS on enhancement of memory, motor learning and neuroplasticity also suggest a role for treatment of cognitive disorders, stroke, and other conditions. The cholinergic activity of the efferent branch of the vagus nerve has an immune inflammatory regulatory effect, which is referred to as the cholinergic anti-inflammatory pathway (CAP).

Upper limb impairment is a frequent outcome of stroke, greatly affecting a patient's quality of life. Recent research has shown that vagus nerve stimulation (VNS) combined with rehabilitation significantly enhances forelimb strength and movement speed in rat models of ischemic stroke. VNS is thought to amplify the advantages of rehabilitation by fostering neuroplasticity.

While the efficacy of taVNS in enhancing motor recovery post-stroke is well-documented, there is a paucity of comparative studies investigating the distinct effects of auricular and cervical tVNS on upper limb function, cognitive outcomes, and quality of life in subacute stroke patients. This gap necessitates further research to determine optimal stimulation modalities and their broader neurorehabilitation benefits

ELIGIBILITY:
Inclusion Criteria:

* First ever ischemic stroke
* Subacute phase of stroke 3-6 months post onset
* Fugl-Meyer Assessment-Upper Extremity (FMA-UE) scores ranged from 20 - 50

Exclusion Criteria:

* Previous injury or surgical intervention of vagus nerve
* Patients with cardiac arrest and arrythmias
* Uncontrolled hypertension
* Apraxia
* Other neurologic or musculoskeletal diseases
* Presence of implanted electronic devices

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Fugl-meyer assessment of upper limb (FMA-UE) | baseline, after 4 weeks, after 8 weeks
  The Fugl-Meyer Assessment-Upper Extremity (FMA-UE) is a commonly utilized tool for measuring motor impairment in stroke rehabilitation. The FMA-UE has demonstrated excellent test-retest and inter- and intra-rater reliability, and evidence for its content validity in acute and subacute populations has been widely reported. The UE section of the FMA consists of 33 items and is scored on a 3-point ordinal scale with 0 meaning cannot perform, 1 meaning can partially perform, and 2 meaning can perform fully. Scores are summed with a maximum potential score of 66 points.
Montreal cognitive assessment (MoCA) | baseline, after 4 weeks, after 8 weeks
  The Montreal Cognitive Assessment (MoCA) is a one-page, 30-point cognitive screening measurement scale that takes about 10 minutes to administer. There are 12 subtasks in the MoCA test that include memory, visuospatial orientation, executive functioning, phonemic fluency, and two-item abstract thinking task, attention, concentration, and working memory, language, orientation to time and place. A score of 26 is a cutoff score to differentiate between normal and abnormal. These findings suggest that MoCA is a reliable and valid tool for detecting major neurocognitive disorders in older populations.
Wolf Motor Function Test (WMFT) | baseline, after 4 weeks, after 8 weeks
  The Wolf Motor Function Test (WMFT) is a standardized assessment tool designed to evaluate upper extremity motor function in individuals who have suffered a stroke or other neurological impairments. It measures the ability to perform tasks that require reaching, grasping, and manipulating objects, focusing on both speed and quality of movement. It is a 21 items scale, ranging from simple movements to more complex actions, allowing for a comprehensive evaluation of motor skills. The items are rated on a 6-point scale, it took approximately 30 minutes.

SECONDARY OUTCOMES:
Stroke-Specific Quality of Life Scale (SS-QOL) | baseline, after 4 weeks, after 8 weeks
  The Stroke-Specific Quality of Life Scale (SS-QOL) is a comprehensive, self-report measure designed specifically to assess health-related quality of life in stroke survivors. The novel 17-item SS-QOL scale (SS-QOL-17) was constructed with the aim of providing a well-balanced measuring tool to depict QOL widely while ensuring the simplicity of administration. It consists of 17- items including mobility, energy, upper extremity function, work/productivity, mood, self-care, social roles, family roles, vision, language, thinking, and personality. Each item is rated on a 5-point Likert scale, with higher scores indicating better function. The total score ranges from 49 to 245, with domain scores calculated as the mean of item scores within each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, Principal Investigator — Lahore University of Biological and Applied Sciences
Locations (1):
- Shadman Medical Center, Stroke Rehabilitation, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hays SA, Rennaker RL, Kilgard MP. Targeting plasticity with vagus nerve stimulation to treat neurological disease. Prog Brain Res. 2013;207:275-99. doi: 10.1016/B978-0-444-63327-9.00010-2. PMID 24309259
- [Background] Hilz MJ. Transcutaneous vagus nerve stimulation - A brief introduction and overview. Auton Neurosci. 2022 Dec;243:103038. doi: 10.1016/j.autneu.2022.103038. Epub 2022 Sep 27. PMID 36201901
- [Background] Butt MF, Albusoda A, Farmer AD, Aziz Q. The anatomical basis for transcutaneous auricular vagus nerve stimulation. J Anat. 2020 Apr;236(4):588-611. doi: 10.1111/joa.13122. Epub 2019 Nov 19. PMID 31742681
- [Background] Murphy SJ, Werring DJ. Stroke: causes and clinical features. Medicine (Abingdon). 2020 Sep;48(9):561-566. doi: 10.1016/j.mpmed.2020.06.002. Epub 2020 Aug 6. PMID 32837228